CLINICAL TRIAL: NCT04387955
Title: Analysis of Chilblains Profile During COVID-19 Epidemic
Brief Title: Analysis of Chilblains pROfile During coVID-19 Epidemic (ACROVID)
Acronym: ACROVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACROVID
Record Dates: First submitted 2020-04-29; First posted 2020-05-14 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: COVID-19; Chilblains
MeSH Terms: conditions — COVID-19; Chilblains

STUDY DESIGN:
Intervention Model Description: Prospective Cohort
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acrovid (Other): Cohort
  Interventions: Diagnostic Test: Biological Sample Collection

INTERVENTIONS:
Diagnostic Test: Biological Sample Collection — * Diagnostic test : biological sample collection at Day 0
  * Two skin biopsies on chilblain at Day 0 (one biopsy for histological analysis, one biopsy for basic research)
  * Anal swabbing at Day 0
  * Blood test at Day 0
  * Blood test at Month 1
  * Blood test at Month 2

SUMMARY:
Cases of chilblains have been reported with an unusual frequency in France in the context of the COronaVirus Infectious Disease 2019 (COVID-19) epidemic. Some of these cases have been linked to a virological status in favour of a recent Severe Acute Respiratory Syndrome CoronaVirus 2 (SARS-CoV-2) infection. Chilblains are acral inflammatory lesion typically reactive to cold (primary form). There are secondary forms acquired during autoimmune connectivitis such as lupus chilblain or hereditary forms related to type I Interferonopathy. An interferon type I signature has been described in these secondary forms of frostbite but also during the cytokine storm of severe forms of CoV-2 SARS infection. If cases of frostbite are indeed secondary to an SARS-CoV-2 infection, comparative analysis of their immunopathological profiles could provide a better understanding of the inflammatory mechanisms during COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of majority or a minor over 12 years of age accompanied by his/her legal representative
* Benefiting from a Social Security scheme
* Informed consent signed by the patient (if major) or by his legal representative (if minor) after clear, fair and appropriate information about the study.
* Red and swollen lesions of the hands and/or feet evolving for more than 24 hours in the context of a COVID-19 epidemic.
* PCR SARS-CoV-2 PCR on nasopharyngeal swab with results available, prior to the inclusion visit.
* Absence of fever or respiratory signs suggestive of COVID-19 for at least 14 days

Exclusion Criteria:

* A person who does not benefit from a Social Security scheme or who does not benefit from it through a third party.
* Patient who is subject to a judicial safeguard measure
* Allergy to local anaesthetic products
* Fever or respiratory signs suggestive of COVID-19 within 14 days

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Study of the link between SARS-CoV-2 infection and chilblains observed during COVID-19 epidemics. | 2 months
  Main Judgement Criterion Comparison between the proportion of patients with chilblains presenting a SARS-CoV-2 positive virological status and the estimated proportion of SARS-CoV-2 positive virological status in the general population.
  The SARS-CoV-2 positive virological status of patients with chilblains will be defined by :
  * SARS-CoV-2 Reverse Transcription-Polymerase Chain Reaction (RT-PCR) on a positive nasopharyngeal swab pre-inclusion.
  * And/or RT-PCR SARS-CoV-2 on positive anal swab at D0
  * And/or RT-PCR SARS-CoV-2 on skin bubble fluid positive at D0.
  * And/or RT-PCR SARS-CoV-2 on skin biopsy positive at D0.
  * And/or SARS-CoV-2 serology positive at D0 and/or M1 and/or M2.

SECONDARY OUTCOMES:
Study of the SARS-CoV-2 virological profile of patients presenting chilblains during a COVID-19 epidemic. | 2 months
  SARS-CoV-2 virological profile of patients with chilblains during a COVID-19 epidemic:
  * Proportion of patients with positive SARS-CoV-2 RT-PCR on pre-inclusion nasopharyngeal swab.
  * Proportion of patients with a positive RT-PCR SARS-CoV-2 on anal self-sampling at D0 +/- M1.
  * Proportion of patients with positive RT-PCR SARS-CoV-2 on skin bubble fluid collection at D0 +/- M1.
  * Proportion of patients with positive RT-PCR SARS-CoV-2 on skin biopsy at D0 and viral quantification.
  * Proportion of patients with positive SARS-CoV-2 serology at D0 and/or M1 and/or M2.
  * Proportion of SARS-CoV-2 positive serum neutralization in patients with SARS-CoV-2 positive serology at D0 and/or M1 and/or M2.
  * Proportion of patients with a positive viral culture at sites with positive PCR (nasopharyngeal or anal or bubble fluid or skin biopsy).
Comparison of the clinical and biological profiles of patients presenting chilblains according to their SARS-CoV-2 virological status (in case of over-representation of SARS-CoV-2 positive patients, the results will be given without comparison). | 2 months
  Comparison between patients with chilblains with a positive SARS-CoV-2 status and patients with chilblains with a negative SARS-CoV-2 status (if there is an overrepresentation of SARS-CoV-2 positive patients, the results will be given without comparison):
  * Proportions of each of the clinical signs detailed in the ACROVID data collection sheet in the Appendix.
  * Proportions of each of the biological characteristics detailed in the ACROVID data collection form in the Appendix.
Comparison of the capillaroscopic profiles of patients with chilblains according to their SARS-CoV-2 virological status (in case of overrepresentation of SARS-CoV-2 positive patients, the results will be given without comparison). | 2 months
  Comparison between patients with chilblains with a positive SARS-CoV-2 status and patients with chilblains with a negative SARS-CoV-2 status (if there is an overrepresentation of SARS-CoV-2 positive patients, the results will be given without comparison):
  - Proportions of each capillaroscopic abnormalities detailed in the ACROVID data collection sheet in the Appendix present during video capillaroscopy performed on all patient fingers (excluding thumbs) at D0 and M2.
Comparison of the TCPO2 profiles of patients with chilblains according to their SARS-CoV-2 virological status (in case of overrepresentation of SARS-CoV-2 positive patients, the results will be given without comparison). | 2 months
  Comparison between patients with chilblains with a positive SARS-CoV-2 status and patients with chilblains with a negative SARS-CoV-2 status (if there is an overrepresentation of SARS-CoV-2 positive patients, the results will be given without comparison):
  - Measurements of TCPO2 (expressed in mmHg) on the inter-metatarsal or metacarpal space of the two most affected toes or fingers.
Comparison of the toe or Finger Pressure Index profiles of patients with chilblains according to their SARS-CoV-2 virological status (in case of overrepresentation of SARS-CoV-2 positive patients, the results will be given without comparison). | 2 months
  Comparison between patients with chilblains with a positive SARS-CoV-2 status and patients with chilblains with a negative SARS-CoV-2 status (if there is an overrepresentation of SARS-CoV-2 positive patients, the results will be given without comparison):
  - Measurements of the toe or finger pressure index calculated as the ratio of the systolic toe or finger pressure measured on the most affected toe or finger (expressed in mmHg) and the average of the humeral systolic arterial pressure (SAP) measured per cuff on both arms (expressed in mmHg).
Comparison of histo-pathological profiles of chilblains according to their SARS-CoV-2 virological status of patients with the disease (in case of overrepresentation of SARS-CoV-2 positive patients, results will be given without comparison). | 2 months
  Comparison between patients with chilblains with a positive SARS-CoV-2 status and patients with chilblains with a negative SARS-CoV-2 status (if there is an overrepresentation of SARS-CoV-2 positive patients, the results will be given without comparison):
  - Proportions of the histological characteristics of skin lesions detailed in the ACROVID data collection form in Appendix COVID-19
Comparison of the gene expression profiles of chilblains according to their SARS-CoV-2 virological status and in healthy subjects. | 2 months
  Comparison between patients with chilblains with a positive SARS-CoV-2 status and patients with chilblains with a negative SARS-CoV-2 status and healthy subjects :
  - Levels of messenger RiboNucleic Acid (mRNA) expression encoding cytokines, chemokines and interferon-induced genes involved in anti-viral response and inflammation in chilblains and Peripheral Blood Mononuclear Cell (PBMC) cultures.
Comparison of the immunostaining profiles of chilblains according to their SARS-CoV-2 virological status and in healthy subjects. | 2 months
  Comparison between patients with chilblains with a positive SARS-CoV-2 status and patients with chilblains with a negative SARS-CoV-2 status and healthy subjects :
  - Immunostaining profiles (qualitative) of cytokines, chemokines and interferon-induced proteins involved in anti-viral response and inflammation in chilblains biopsy sections.
Comparison of the ELISA assays profiles of chilblains according to their SARS-CoV-2 virological status and in healthy subjects. | 2 months
  Comparison between patients with chilblains with a positive SARS-CoV-2 status and patients with chilblains with a negative SARS-CoV-2 status and healthy subjects :
  - ELISA assays of cytokines and chemokines involved in anti-viral response and inflammation in plasma and PBMC supernatant from patients with chilblains.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France